CLINICAL TRIAL: NCT04669509
Title: Effect of Liver Injury on Mortality in Coronavirus Disease-2019 Patients Admitted to Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cem Kıvılcım Kaçar, Anesthesiology and reanimation specialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: CKKacar
Record Dates: First submitted 2020-12-14; First posted 2020-12-16 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Covid19; Liver Injury; Mortality
MeSH Terms: conditions — COVID-19 | interventions — Liver Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with normal ALT, AST and total bilirubin values
  Interventions: Diagnostic Test: Liver function tests
- Group 2: Patients whose ALT, AST or total bilirubin levels are up to 3 times upper limit of normal
  Interventions: Diagnostic Test: Liver function tests
- Group 3: Patients whose ALT, AST or total bilirubin levels are increased more than 3 times upper limit of normal
  Interventions: Diagnostic Test: Liver function tests

INTERVENTIONS:
Diagnostic Test: Liver function tests — Patients' age, gender, comorbidity, Acute Physiology and Chronic Health Evaluation II (APACHE II), Sequential Organ Failure Assessment (SOFA) scores when first admitted to the ICU, hemogram parameters (white blood cell count, neutrophil, lymphocyte, hemoglobin, platelet count), coagulation parameters (prothrombin time, activated partial thromboplastin time and D-dimer, blood biochemistry results (C-reactive protein, lactate dehydrogenase, creatine kinase , alanine aminotransferase, aspartate aminotransferase, total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded. It will also be recorded whether mortality develops on day 7 and day 28.

SUMMARY:
In addition to primarily affecting the lungs, coronavirus disease-2019 (COVID-19) disease can also affect many different organs, especially the heart, kidneys, liver and brain. In this group of patients, the impact of an important organ such as the liver can lead to a further deterioration of the clinical course. In this study, critical patients admitted to Gazi Yasargil Training and Research Hospital intensive care unit (ICU) due to COVID-19 between April 1 and October 1, 2020 were retrospectively analyzed. The effect of liver damage on mortality in critical COVID-19 patients was investigated. The necessary permits for the study were obtained from the Scientific Research Platform of the T.R. Ministry of Health. (20.11.2020) Patients diagnosed with COVID-19 on the specified dates, followed in the ICU, older than 18 years, identified as critical/serious according to the World Health Organization and provisional guidelines of the Scientific Board of the T.R. Ministry of Health will be included in the study.

ICU patients without COVID-19, COVID-19 patients under 18 years of age,COVID-19 patients with known liver disease, and COVID-19 patients with mild to moderate symptoms will be excluded from the study.

Patients' age, gender, comorbidity, Acute Physiology and Chronic Health Evaluation II (APACHE II), Sequential Organ Failure Assessment (SOFA) scores when first admitted to the ICU, hemogram parameters (white blood cell count, neutrophil, lymphocyte, hemoglobin, platelet count), coagulation parameters (prothrombin time, activated partial thromboplastin time and D-dimer, blood biochemistry results (C-reactive protein, lactate dehydrogenase, creatine kinase , alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, direct bilirubin and indirect bilirubin), procalcitonin and ferritin levels will be recorded. In addition, the number of days spent in the ICU and whether mortality develops or not will be recorded. It will also be recorded whether mortality develops on day 7 and day 28.

Patients will be divided into three groups according to their ALT, AST and total bilirubin levels at the time of admission to the ICU. Group 1 will consist of patients with normal ALT, AST and total bilirubin values. Group 2 will consist of patients whose ALT, AST or total bilirubin levels are up to 3 times upper limit of normal. Group 3 will consist of patients whose ALT, AST or total bilirubin levels are increased more than 3 times upper limit of normal.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19 on the specified dates, followed in the ICU, older than 18 years, identified as critical/serious according to the World Health Organization and provisional guidelines of the Scientific Board of the T.R. Ministry of Health will be included in the study.

Exclusion Criteria:

* ICU patients without COVID-19, COVID-19 patients under 18 years of age,COVID-19 patients with known liver disease, and COVID-19 patients with mild to moderate symptoms will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients admitted to Gazi Yasargil Training and Research Hospital intensive care unit (ICU) due to COVID-19 between April 1 and October 1, 2020
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
7 and 28 day mortality | Patients hospitalized in the ICU within 6 months
  Effect of Liver Injury on Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cai Q, Huang D, Yu H, Zhu Z, Xia Z, Su Y, Li Z, Zhou G, Gou J, Qu J, Sun Y, Liu Y, He Q, Chen J, Liu L, Xu L. COVID-19: Abnormal liver function tests. J Hepatol. 2020 Sep;73(3):566-574. doi: 10.1016/j.jhep.2020.04.006. Epub 2020 Apr 13. PMID 32298767
- [Background] Huang H, Chen S, Li H, Zhou XL, Dai Y, Wu J, Zhang J, Shao L, Yan R, Wang M, Wang J, Tu Y, Ge M. The association between markers of liver injury and clinical outcomes in patients with COVID-19 in Wuhan. Aliment Pharmacol Ther. 2020 Sep;52(6):1051-1059. doi: 10.1111/apt.15962. Epub 2020 Jul 22. PMID 32697870
- [Background] Jiang S, Wang R, Li L, Hong D, Ru R, Rao Y, Miao J, Chen N, Wu X, Ye Z, Hu Y, Xie M, Zuo M, Lu X, Qiu Y, Liang T. Liver Injury in Critically Ill and Non-critically Ill COVID-19 Patients: A Multicenter, Retrospective, Observational Study. Front Med (Lausanne). 2020 Jun 23;7:347. doi: 10.3389/fmed.2020.00347. eCollection 2020. PMID 32656222
- [Background] Fan Z, Chen L, Li J, Cheng X, Yang J, Tian C, Zhang Y, Huang S, Liu Z, Cheng J. Clinical Features of COVID-19-Related Liver Functional Abnormality. Clin Gastroenterol Hepatol. 2020 Jun;18(7):1561-1566. doi: 10.1016/j.cgh.2020.04.002. Epub 2020 Apr 10. PMID 32283325